CLINICAL TRIAL: NCT00738829
Title: Fludarabine/Rituximab Combined With Escalating Doses of Lenalidomide Followed by Rituximab/Lenalidomide in Untreated Chronic Lymphocytic Leukemia (CLL) - a Dose-finding Study With Concomitant Evaluation of Safety and Efficacy.
Brief Title: Lenalidomide Dose Escalation Combined With Rituximab/Fludarabine in Untreated CLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Celgene Corporation (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL-5; EudraCT Nr. 2008-001430-27; ML21718
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: CLL; untreated; immune therapy; dose escalation; maximum tolerated dose; maintenance therapy; Lenalidomide; Rituximab; Fludarabine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; fludarabine; fludarabine phosphate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Lenalidomide Dose Escalation combined with Fludarabine/Rituximab followed by maximum tolerated lenalidomide dose/Rituximab maintenance therapy
  Interventions: Drug: Lenalidomide; Drug: Fludarabine; Biological: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Dose escalation stage: starting dose 2.5mg/d, dose escalation via 5/10/15/20/25 mg/d every 28 days if no dose-limiting toxicity.
  During maintenance stage dosing on days 1-28 for max. 6 months at maximum tolerated dose reached during dose escalation stage.
  Other Names: Revlimid
Drug: Fludarabine — 25 mg/m2 i.v. d1-3 or 40 mg/m2 po d1-3 every 28 days for 6 cycles during dose escalation stage.
  Other Names: Fludarabine phosphate
Biological: Rituximab — Dose escalation stage: 375 mg/m2 i.v. d4 Cycle 1, 500 mg/m2 i.v. d1 Cycles 2-6.
  Maintenance stage: 375 mg/m2 i.v. at 2/4/6 months after end of escalation stage.
  Other Names: MabThera

SUMMARY:
The aim of this study is to determine the maximal tolerated dose level of lenalidomide combined with fludarabine/rituximab in the therapy of patients with previously untreated CD20-positive chronic lymphocytic leukemia. Following a dose escalation phase lenalidomide will be given at the pre-determined maximum tolerated dose in combination with rituximab to further determine the efficacy and tolerability of this regimen.

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, open-label, single-arm Phase I/II study in patients with previously untreated CD20-positive CLL. Phase I of the study will evaluate the maximal tolerated lenalidomide dose level in combination with fludarabine/rituximab chemoimmunotherapy in 10 patients. Phase II will determine efficacy using the combination in the previously defined maximal tolerated dose. Both phases will be followed by a maintenance phase evaluating the tolerability and possibility to further improve response quality.

ELIGIBILITY:
Inclusion Criteria:

* B-CLL (CD23+, CD5+, CD19+, CD20+)
* Treatment indication according to NCI criteria
* Age >= 18 yrs
* No previous treatment of CLL by chemo-, radio- or immunotherapy
* Life expectancy > 6 months
* Written informed consent
* Women of non-childbearing potential or women of childbearing potential and men using effective contraception

Exclusion Criteria:

* Active bacterial, viral or fungal infection
* Positivity for HIV, Hepatitis B or C
* Reduce organ functions and bone marrow dysfunction not due to CLL
* Creatinine clearance below 30 ml/min
* Patients with medical conditions requiring long-term use of systemic corticosteroids during study treatment
* Patients with a history of severe cardiac disease
* Other known co-morbidity with the potential to dominate survival
* Transformation to aggressive B-cell malignancy
* Known hypersensitivity to humanised monoclonal antibodies or any of the study drugs
* Pregnant or breast-feeding women
* Any co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Lenalidomide Maximum Tolerated Dose | Dose escalation stage

SECONDARY OUTCOMES:
Safety profile of Lenalidomide/Fludarabine/Rituximab treatment | Study Duration
Safety Profile of Lenalidomide/Rituximab | Study duration
Response rate for Lenalidomide/Fludarabine/Rituximab combination treatment | Dose escalation stage
Response rate for Lenalidomide/Rituximab combination therapy | Study Duration
Response rate by 4-colour flow cytometric MRD analysis | Study Duration
Changes in Quality of Life scores | Study Duration
Risk factors and clonal evolution | Study Duration

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, Prof. Dr., Principal Investigator — Universitaetsklinik f. Innere Medizin III, Universitaetsklinikum der PMU, Salzburg
Locations (7):
- Austria (7):
  - Medizinische Universitaet Innsbruck, Abtlg. f. Haematologie und Onkologie, Innsbruck, Tyrol
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Krankenhaus d. Barmherzigen Schwestern Linz, Linz
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Krankenhaus der Stadt Linz, Linz
  - Universitaetsklinik f. Innere Medizin III, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, Wels

REFERENCES:
- [Derived] Egle A, Steurer M, Melchardt T, Weiss L, Gassner FJ, Zaborsky N, Geisberger R, Catakovic K, Hartmann TN, Pleyer L, Voskova D, Thaler J, Lang A, Girschikofsky M, Petzer A, Greil R. Fludarabine and rituximab with escalating doses of lenalidomide followed by lenalidomide/rituximab maintenance in previously untreated chronic lymphocytic leukaemia (CLL): the REVLIRIT CLL-5 AGMT phase I/II study. Ann Hematol. 2018 Oct;97(10):1825-1839. doi: 10.1007/s00277-018-3380-z. Epub 2018 Jun 4. PMID 29862437